CLINICAL TRIAL: NCT05218122
Title: To Explore the Characteristics of LKD Syndrome and PBS Syndrome of Knee Osteoarthritis Which Based on the Enhancement of Inflammatory Response Caused by the Inhibition of TGF-β/Smad Signal Pathway
Brief Title: Characteristics of LKDS and PBSS of KOA Based on the Enhancement of Inflammatory Response by TGF-β/Smad Pathway Inhibited
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Chao Ye, Principal Investigator, Dongzhimen Hospital, Beijing
Other Study IDs: 2021DZMEC-139-03
Record Dates: First submitted 2021-12-27; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Knee Osteoarthritis; Syndrome; Traditional Chinese Medicine
Keywords: TGF-β/Smad signaling pathway; disease and syndrome cell model; knee osteoarthritis; syndrome; traditional Chinese medicine
MeSH Terms: conditions — Osteoarthritis, Knee; Syndrome; Disease | interventions — Cross-Sectional Studies; Methods

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- LKD syndrome: liver and kidney deficiency syndrome
  Interventions: Other: cross-sectional study without intervention
- PBS syndrome: phlegm and blood stasis syndrome
  Interventions: Other: cross-sectional study without intervention
- NC group: Normal Control group
  Interventions: Other: cross-sectional study without intervention

INTERVENTIONS:
Other: cross-sectional study without intervention — cross-sectional study without intervention

SUMMARY:
1. Through research and analysis, the levels of upstream and downstream factors related to TGF-β/Smad signaling pathway and inflammatory response factor related factors in serum, blood cells, articular fluid, urine, tongue covering and discarded tissues after surgery of patients with LKD syndrome and PBS syndrome of knee osteoarthritis were obtained, and the syndrome characteristics were further obtained.
2. Through research and analysis, the index levels of multiple omics detection in serum, blood cells, joint fluid, urine, tongue coating and discarded tissues of patients with LKD syndrome and PBS syndrome of knee osteoarthritis were obtained, and the syndrome characteristics were further obtained.
3. The severity of syndrome was quantified by syndrome score scale and the correlation between the above results and the syndrome score of patients with knee osteoarthritis with LKD syndrome and PBS syndrome was studied in combination with imaging characteristics.
4. To establish a "disease and syndrome cell model" and test relevant indicators to support the above research.
5. Through the analysis of the above research results, the possible mechanism is analyzed to provide an objective basis for the biological basis of the syndrome and relevant evidence for the clinical diagnosis and treatment of knee osteoarthritis with traditional Chinese medicine.

DETAILED DESCRIPTION:
1. Through research and analysis, the levels of upstream and downstream factors related to TGF-β/Smad signaling pathway and inflammatory response factor related factors in serum, blood cells, articular fluid, urine, tongue covering and discarded tissues after surgery of patients with liver and kidney deficiency syndrome and phlegm and blood stasis syndrome of knee osteoarthritis were obtained, and the syndrome characteristics were further obtained.
2. Through research and analysis, the index levels of multiple omics detection in serum, blood cells, joint fluid, urine, tongue coating and discarded tissues of patients with liver and kidney deficiency syndrome and phlegm and blood stasis syndrome of knee osteoarthritis were obtained, and the syndrome characteristics were further obtained.
3. The severity of syndrome was quantified by syndrome score scale and the correlation between the above results and the syndrome score of patients with knee osteoarthritis with liver and kidney deficiency syndrome and phlegm and blood stasis syndrome was studied in combination with imaging characteristics.
4. To establish a "disease and syndrome cell model" and test relevant indicators to support the above research.
5. Through the analysis of the above research results, the possible mechanism is analyzed to provide an objective basis for the biological basis of the syndrome and relevant evidence for the clinical diagnosis and treatment of knee osteoarthritis with traditional Chinese medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria of liver and kidney deficiency syndrome and phlegm and blood stasis syndrome in knee osteoarthritis

   * Age 20-80 years old, in line with the diagnostic criteria of Western medicine;
   * In accordance with the diagnostic criteria of TCM syndromes, it belongs to liver and kidney deficiency syndrome and phlegm and blood stasis syndrome;
   * Patients who are willing to participate in the survey and have good compliance;
   * Voluntary signing of informed consent;
2. Inclusion criteria of normal control group

   * Age 20-80 years old.
   * Patients who are willing to participate in the survey and have good compliance.
   * It does not meet the diagnostic criteria of knee osteoarthritis.
   * Voluntarily sign informed consent.

Exclusion Criteria:

* Complications affecting joints, such as psoriasis, syphilitic neuropathy, brown yellow disease, metabolic bone disease, etc;
* There were rheumatoid arthritis and ankylosing spondylitis;
* Late disabled and incapacitated;
* Pregnant or lactating women;
* Mentally ill.
* As long as one of the above 5 articles is met, it shall be excluded.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Among the outpatients and inpatients in Dongzhimen Hospital of Beijing University of traditional Chinese medicine from December 2021 to August 2024, 150 cases of liver and kidney deficiency syndrome and 300 cases of phlegm and blood stasis syndrome were taken respectively. All patients met the diagnosis of knee osteoarthritis and met the inclusion criteria. Another 40 cases of normal control group were taken.
Sampling Method: Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2021-12-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
the differences of metabonomics | 3 years
  The differences of metabonomics in blood, urine and tongue coating will be detected by metabonomics in LKD group, PBS group and NC group.
the differences of metabonomics in the cell models of disease-TCM syndrome | 3 years
  The differences of metabonomics in the cell models of disease-TCM syndrome will be detected by metabonomics.
the differences of proteomics in the cell models of disease-TCM syndrome | 3 years
  The differences of proteomics in the cell models of disease-TCM syndrome will be detected by proteomics.
the differences of proteomics | 3 years
  The differences of proteomics in blood, urine and tongue coating will be detected by proteomics in LKD group, PBS group and NC group.
the differences of transcriptomics | 3 years
  The differences of transcriptomics in blood, urine and tongue coating will be detected by transcriptomics in LKD group, PBS group and NC group.
the differences of transcriptomics in the cell models of disease-TCM syndrome | 3 years
  The differences of transcriptomics in the cell models of disease-TCM syndrome will be detected by transcriptomics.
the related indexes of TGF- β/ Smad signaling pathway and inflammatory response | 3 years
  Histological and pathological examination is used to detect the related indexes of TGF- β/ Smad signaling pathway and inflammatory response.
The clinical TCM scores of LKD | 3 years
  The minimum value is 0 and maximum value is 38, and higher scores mean a worse outcome.
The clinical TCM scores of PBS | 3 years
  The minimum value is 0 and maximum value is 41, and higher scores mean a worse outcome.
The grading scores of Kellgren Lawrence (K-L) | 3 years
  The minimum value is 0 and maximum value is 4, and higher scores mean a worse outcome.
The grading scores of Yulish | 3 years
  The minimum value is 0 and maximum value is 4, and higher scores mean a worse outcome.
Clinical data | 3 years
  Collect clinical data and formulate a unified questionnaire, including the name, age, gender, outpatient / inpatient number, past history, current medical history, imaging images and other relevant data of patients with knee osteoarthritis.
Concentration of BLC (CXCL13) | 3 years
  Concentration of BLC (CXCL13) will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of BLC (CXCL13) in the cell models of disease-TCM syndrome | 3 years
  Concentration of BLC (CXCL13) will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of Eotaxin-1 (CCL11) | 3 years
  Concentration of Eotaxin-1 (CCL11) will be detected by ELISA will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of Eotaxin-1 (CCL11) in the cell models of disease-TCM syndrome | 3 years
  Concentration of Eotaxin-1 (CCL11) will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of Eotaxin-2 (MPIF-2/CCL24) | 3 years
  Concentration of Eotaxin-2 (MPIF-2/CCL24) will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of Eotaxin-2 (MPIF-2/CCL24) in the cell models of disease-TCM syndrome | 3 years
  Concentration of Eotaxin-2 (MPIF-2/CCL24) will be detected by ELISA in the cell models of disease-TCM.
Concentration of GCSF | 3 years
  Concentration of GCSF will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of GCSF in the cell models of disease-TCM syndrome | 3 years
  Concentration of GCSF will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of GM-CSF | 3 years
  Concentration of GM-CSF will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of GM-CSF in the cell models of disease-TCM syndrome | 3 years
  Concentration of GM-CSF will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of I-309 (TCA-3/CCL1) | 3 years
  Concentration of I-309 (TCA-3/CCL1) will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of I-309 (TCA-3/CCL1) in the cell models of disease-TCM syndrome | 3 years
  Concentration of I-309 (TCA-3/CCL1) will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of ICAM-1(CD54) | 3 years
  Concentration of ICAM-1(CD54) will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of ICAM-1(CD54) in the cell models of disease-TCM syndrome | 3 years
  Concentration of ICAM-1(CD54) will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of IFN-gamma | 3 years
  Concentration of IFN-gamma will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of IFN-gamma in the cell models of disease-TCM syndrome | 3 years
  Concentration of IFN-gamma will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of IL-1 alpha (IL-1 F1) | 3 years
  Concentration of IL-1 alpha (IL-1 F1) will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of IL-1 alpha (IL-1 F1) in the cell models of disease-TCM syndrome | 3 years
  Concentration of IL-1 alpha (IL-1 F1) will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of IL-1 beta (IL-1 F2) | 3 years
  Concentration of IL-1 beta (IL-1 F2) will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of IL-1 beta (IL-1 F2) in the cell models of disease-TCM syndrome | 3 years
  Concentration of IL-1 beta (IL-1 F2) will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of IL-1 ra (IL-1 F3) | 3 years
  Concentration of IL-1 ra (IL-1 F3) will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of IL-1 ra (IL-1 F3) in the cell models of disease-TCM syndrome | 3 years
  Concentration of IL-1 ra (IL-1 F3) will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of IL-2 | 3 years
  Concentration of IL-2 will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of IL-2 in the cell models of disease-TCM syndrome | 3 years
  Concentration of IL-2 will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of IL-4 | 3 years
  Concentration of IL-4 will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of IL-4 in the cell models of disease-TCM syndrome | 3 years
  Concentration of IL-4 will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of IL-5 | 3 years
  Concentration of IL-5 will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of IL-5 in the cell models of disease-TCM syndrome | 3 years
  Concentration of IL-5 will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of IL-6 | 3 years
  Concentration of IL-6 will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of IL-6 in the cell models of disease-TCM syndrome | 3 years
  Concentration of IL-6 will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of IL-6R | 3 years
  Concentration of IL-6R will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of IL-6R in the cell models of disease-TCM syndrome | 3 years
  Concentration of IL-6R will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of IL-7 | 3 years
  Concentration of IL-7 will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of IL-7 in the cell models of disease-TCM syndrome | 3 years
  Concentration of IL-7 will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of IL-8(CXCL8) | 3 years
  Concentration of IL-8(CXCL8) will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of IL-8(CXCL8) in the cell models of disease-TCM syndrome | 3 years
  Concentration of IL-8(CXCL8) will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of IL-10 | 3 years
  Concentration of IL-10 will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of IL-10 in the cell models of disease-TCM syndrome | 3 years
  Concentration of IL-10 will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of IL-11 | 3 years
  Concentration of IL-11 will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of IL-11 in the cell models of disease-TCM syndrome | 3 years
  Concentration of IL-11 will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of IL-12 p40 | 3 years
  Concentration of IL-12 p40 will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of IL-12 p40 in the cell models of disease-TCM syndrome | 3 years
  Concentration of IL-12 p40 will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of IL-12 p70 | 3 years
  Concentration of IL-12 p70 will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of IL-12 p70 in the cell models of disease-TCM syndrome | 3 years
  Concentration of IL-12 p70 will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of IL-13 | 3 years
  Concentration of IL-13 will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of IL-13 in the cell models of disease-TCM syndrome | 3 years
  Concentration of IL-13 will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of IL-15 | 3 years
  Concentration of IL-15 will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of IL-15 in the cell models of disease-TCM syndrome | 3 years
  Concentration of IL-15 will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of IL-16 | 3 years
  Concentration of IL-16 will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of IL-16 in the cell models of disease-TCM syndrome | 3 years
  Concentration of IL-16 will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of IL-17A | 3 years
  Concentration of IL-17A will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of IL-17A in the cell models of disease-TCM syndrome | 3 years
  Concentration of IL-17A will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of MCP-1 (CCL2) | 3 years
  Concentration of MCP-1 (CCL2) will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of MCP-1 (CCL2) in the cell models of disease-TCM syndrome | 3 years
  Concentration of MCP-1 (CCL2) will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of M-CSF | 3 years
  Concentration of M-CSF will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of M-CSF in the cell models of disease-TCM syndrome | 3 years
  Concentration of M-CSF will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of MIG (CXCL9) | 3 years
  Concentration of MIG (CXCL9) will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of MIG (CXCL9) in the cell models of disease-TCM syndrome | 3 years
  Concentration of MIG (CXCL9) will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of MIP-1 | 3 years
  Concentration of MIP-1 will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of MIP-1 in the cell models of disease-TCM syndrome | 3 years
  Concentration of MIP-1 will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of alpha (CCL3) in the cell models of disease-TCM syndrome | 3 years
  Concentration of alpha (CCL3) will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of alpha (CCL3) | 3 years
  Concentration of alpha (CCL3) will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of MIP-1 beta (CCL4) | 3 years
  Concentration of MIP-1 beta (CCL4) will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of MIP-1 beta (CCL4) in the cell models of disease-TCM syndrome | 3 years
  Concentration of MIP-1 beta (CCL4) will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of MIP-1 delta (CCL15) | 3 years
  Concentration of MIP-1 delta (CCL15) will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of MIP-1 delta (CCL15) in the cell models of disease-TCM syndrome | 3 years
  Concentration of MIP-1 delta (CCL15) will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of PDGF-BB | 3 years
  Concentration of PDGF-BB will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of PDGF-BB in the cell models of disease-TCM syndrome | 3 years
  Concentration of PDGF-BB will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of RANTES (CCL5) | 3 years
  Concentration of RANTES (CCL5) will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of RANTES (CCL5) in the cell models of disease-TCM syndrome | 3 years
  Concentration of RANTES (CCL5) will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of TIMP-1 | 3 years
  Concentration of TIMP-1 will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of TIMP-1 in the cell models of disease-TCM syndrome | 3 years
  Concentration of TIMP-1 will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of TIMP-2 | 3 years
  Concentration of TIMP-2 will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of TIMP-2 in the cell models of disease-TCM syndrome | 3 years
  Concentration of TIMP-2 will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of TNF alpha | 3 years
  Concentration of TNF alpha will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of TNF alpha in the cell models of disease-TCM syndrome | 3 years
  Concentration of TNF alpha will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of TNF beta (TNFSF1B) | 3 years
  Concentration of TNF beta (TNFSF1B) will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of TNF beta (TNFSF1B) in the cell models of disease-TCM syndrome | 3 years
  Concentration of TNF beta (TNFSF1B) will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of TNF RI (TNFRSF1A) | 3 years
  Concentration of TNF RI (TNFRSF1A) will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of TNF RI (TNFRSF1A) in the cell models of disease-TCM syndrome | 3 years
  Concentration of TNF RI (TNFRSF1A) will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of TNF RII(TNFRSF1B) | 3 years
  Concentration of TNF RII(TNFRSF1B) will be detected by ELISA in LKD group, PBS group and NC group.
Concentration of TNF RII(TNFRSF1B) in the cell models of disease-TCM syndrome | 3 years
  Concentration of TNF RII(TNFRSF1B) will be detected by ELISA in the cell models of disease-TCM syndrome.
Concentration of Signaling pathway indicator | 3 years
  Concentration of Signaling pathway indicator will be detected by ELISA, metabonomics, proteomics, transcriptomics in LKD group, PBS group and NC group.
Concentration of Signaling pathway indicator in the cell models of disease-TCM syndrome | 3 years
  Concentration of Signaling pathway indicator will be detected by ELISA, metabonomics, proteomics, transcriptomics in the cell models of disease-TCM syndrome.
Concentration of Routine Blood Examination （Concentration of WBC, LYMPH%, MONO, NEUT%, LYMPH, MONO%, NEUT, BASO%, BASO, MCH, MCHC,ROW-CV, MPV, PLT, PDW, EO%, P-LCR, RBC, Hb, HCT） | 3 years
  LKD group, PBS group and NC group's Routine Blood Examination will be detect by automated hematology analyzer.
Concentration of Blood Biochemistry (Concentration of TC, TG, HDL-C, LDL-C, Urea, Cr, UA, GLu, ALT, AST, TP, ALB, ALP, GGT, TBIL, DBIL, Mg, K, Na, Cl, Ca, P, Fe, CO2) | 3 years
  LKD group, PBS group and NC group's Blood Biochemistry will be detect by automatic biochemical analyzer.
Concentration of Routine Urine Examination (Concentration of LEU, NIT, PRO, GLU-U, KET, URO, BIL, PH-U, SG, BLU) | 3 years
  LKD group, PBS group and NC group's Routine Urine Examination will be detect by Urine analyzer.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongzhimen Hospital, Beijing, Beijing Municipality, China